CLINICAL TRIAL: NCT01881932
Title: Acupuncture to Prevent Chemotherapy Dose Reduction Due to Chemotherapy-induced Peripheral Neuropathy in Breast and Colorectal Cancer Patients
Brief Title: Acupuncture to Prevent Chemotherapy Dose Reduction Due to Chemotherapy-induced Peripheral Neuropathy in Breast and Colorectal Cancer Patients (GCC1232)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has moved to another institution, which resulted in significant changes in the study design and study title.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HP-00053394; GCC1232 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2013-03-13; First posted 2013-06-20 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: acupuncture therapy; sham acupuncture therapy; chemotherapy-induced peripheral neuropathy (CIPN)
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (No Intervention): Patients will be stratified based on cancer type (breast cancer vs colorectal cancer). In standard care arm, patients will not receive additional therapy for CIPN. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemotherapy received in the past week. Record how much chemotherapy received all together. Each week patient will have blood drawn (about 1 teaspoon) to check nerve growth factors levels. All patients will follow the same chemotherapy dose reduction algorithm. No concomitant anti-neuropathy medication is allowed.
- Acupuncture (Experimental): Patients will be stratified based on cancer type (breast cancer vs colorectal cancer). The patients will be randomly assigned to receive acupuncture until the end of their chemotherapy. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemotherapy received in the past week. Record how much chemotherapy received all together. Each week patient will have blood drawn (about 1 teaspoon) to check nerve growth factors levels. All patients will follow the same chemotherapy dose reduction algorithm. No concomitant anti-neuropathy medication is allowed. In standard care arm, patients will not receive additional therapy for CIPN.
  Interventions: Device: Acupuncture using Seirin® needles
- Sham Acupuncture (Active Comparator): Patients will be stratified based on cancer type (breast cancer vs colorectal cancer). The patients will be randomly assigned to receive sham acupuncture until the end of their chemotherapy while following the same chemotherapy dose reduction algorithm. No concomitant anti-neuropathy medication is allowed. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemotherapy received in the past week. Record how much chemotherapy received all together. Each week patient will have blood drawn (about 1 teaspoon) to check nerve growth factors levels.
  Interventions: Device: Sham Acupuncture using Park Sham placebo acupuncture device

INTERVENTIONS:
Device: Acupuncture using Seirin® needles — Participants will receive acupuncture weekly until the end of chemotherapy.
  Subjects will receive acupuncture at documented acupoints. To improve blinding effect, the acupuncturist will also tap 2 guiding tubes at 2 sham points , and immediately affix a pair of needles to the surface of the same points with adhesive tape, without needle insertion.
  Arms: Acupuncture
Device: Sham Acupuncture using Park Sham placebo acupuncture device — Participants will receive sham acupuncture until the end of chemotherapy.
  Acupuncturist will insert Park Sham Devices, non-penetrating sham acupuncture device consisting of a retractable needle and an adhesive tube into the sham points, and then immediately apply 2 pieces of adhesive tape next to the needles. In addition, she will tap a mock plastic needle guiding tube on the surface of each of the 8 true points in the arm and leg to produce some discernible sensation and then immediately apply a needle with a piece of adhesive tape to the dermal surface, without needle insertion.
  Arms: Sham Acupuncture

SUMMARY:
In this study the investigators will assess how useful and safe acupuncture is in easing the pain, tingling and numbness that is caused by chemotherapy. The researchers hope this will prevent the need to reduce the amount of chemotherapy a patient receives.

DETAILED DESCRIPTION:
This is a single-center, pilot (phase IIb), randomized, standard care- and placebo (sham acupuncture)-controlled clinical trial (N=60) assessing the effects of acupuncture to prevent chemotherapy dose reduction due to chemotherapy-induced peripheral neuropathy (CIPN) and to elucidate the mechanism of action. Breast or colorectal cancer patients receiving neoadjuvant or adjuvant chemotherapy containing neurotoxic agents (taxanes or oxaliplatin) at the University of Maryland Marlene & Stewart Greenebaum Cancer Center (UMGCC) will be screened for CIPN. Once these patients develop greater than or equal to National Cancer Institute-Common Toxicity Criteria (NCI-CTC) grade 2 CIPN, they will be recruited for this study. Severity of CIPN as defined by NCI-CTC is listed in Appendix A. Patients will be stratified based on cancer type (breast cancer vs colorectal cancer). The patients will then be randomly assigned to one of three arms: (A) real acupuncture, (B) sham acupuncture or (C) standard care. All patients will follow the same chemotherapy dose reduction algorithm (Appendix B). No concomitant anti-neuropathy medication is allowed. Patients in the intervention arms will be randomly assigned to undergo weekly real or sham acupuncture until the end of their chemotherapy. In these two arms, the patient, the patient's medical oncologist, pharmacist, research nurse, and study coordinator will be blinded to the treatment assignment. In standard care arm, patients will not receive additional therapy for CIPN. Their CIPN will be managed according to the standard chemotherapy dose reduction algorithm. In all arms, chemotherapy dose will be documented during the patient's scheduled chemotherapy sessions. The chemotherapy relative dose intensity (RDI) will be calculated at the end of their chemotherapy. Validated patient-reported outcome questionnaires: Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) questionnaire and Neuropathy Pain Scale (NPS), described later, will be used to assess CIPN severity weekly in all patients until the end of their chemotherapy and at the 4 week follow up. Nerve conduction study will be performed by a neurologist at baseline and after chemotherapy is finished. Side effects from real or sham acupuncture will be recorded weekly. Approximately 4 ml of blood will be drawn from patients before each real or sham acupuncture treatment, or with routine weekly blood work check (in the standard care arm), at the end of chemotherapy, and at the 4 week follow up to measure changes in nerve growth factor and other neurotrophic factors such as brain-derived neurotrophic factor, neurotrophin-3, the insulin-like growth factors, and vascular endothelial growth factor. They will be analyzed in the cytokine lab at the University of Maryland School of Medicine (UMSOM).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage I-III carcinoma of the breast OR histologically proven stage I-III colorectal carcinoma.
* Receiving adjuvant or neoadjuvant chemotherapy that includes a taxane or oxaliplatin.
* While on chemotherapy, develop greater than or equal to NCI-CTC grade 2 CIPN.
* Eastern Cooperative Oncology Group performance status 0-2.
* The patient is aware of the nature of his/her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Prior acupuncture within one year of enrollment.
* Known metastatic (stage IV) breast or colorectal cancer involvement.
* Pre-existing peripheral neuropathy before chemotherapy is initiated
* Currently taking anti-neuropathy medication such as gabapentin, or pregabalin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, DABMA, Principal Investigator — University of Maryland Marlene & Stewart Greenebaum Cancer Center
Locations (1):
- University of Maryland Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University Medical Centers and Hospital Based Oncology Programs recruited participants from February 2013 until June 2014.
Pre-assignment Details: Nineteen patients were enrolled and randomly assigned to one of three arms: a) real acupuncture, b) sham acupuncture or c) standard of care. Two patients received standard of care, 4 real and 13 sham.
Groups:
- Acupuncture: Patients will be stratified based on cancer type (breast cancer vs colorectal cancer). Patients will be randomly assigned to receive acupuncture until the end of their chemotherapy. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemotherapy received in the past week. Record how much chemotherapy received all together. Each week patient will have blood drawn (about 1 teaspoon) to check nerve growth factors levels. All patients will follow the same chemotherapy dose reduction algorithm. No concomitant anti-neuropathy medication is allowed. In standard care arm, patients will not receive additional therapy for CIPN.
  Acupuncture using Seirin® needles: Participants will receive acupuncture weekly until the end of chemotherapy.
  Subjects will receive acupuncture at documented acupoints. To improve blinding effect, the acupuncturist will also tap 2 guiding tubes at 2 sham points, and
- Sham Acupuncture: Patients will be stratified based on cancer type (breast cancer vs colorectal cancer). The patients will be randomly assigned to receive sham acupuncture until the end of their chemotherapy while following the same chemotherapy dose reduction algorithm. No concomitant anti-neuropathy medication allowed. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemotherapy received in the past week. Record how much chemotherapy received all together. Each week patient will have blood drawn (about 1 teaspoon) to check nerve growth factors levels.
  Sham Acupuncture using Park Sham placebo acupuncture device: Participants will receive sham acupuncture until the end of chemotherapy.
  Acupuncturist will insert Park Sham Devices, non-penetrating sham acupuncture device consisting of a retractable needle and an adhesive tube into the sham points, and then immediately apply 2 pieces of adhesive tape
Period: Overall Study
Arm/Group | Standard Care | Acupuncture | Sham Acupuncture
Started | 2 | 4 | 13
Completed | 2 | 4 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acupuncture: Pts stratified based on cancer (breast cancer vs colorectal cancer). Patients randomly assigned to get acupuncture until the end of their chemo. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemo received in past week. Record how much chemo received all together. Each week patient will have blood drawn (about 1 tsp) to check nerve growth factors levels. All patients will follow the same chemo dose reduction algorithm. No concomitant anti-neuropathy medication allowed. In standard care arm, patients will not get addiinl therapy for CIPN. Acupuncture using Seirin® needles: Participants will get acupuncture weekly til the end of chemo. Subjects will receive acupuncture at documented acupoints. To improve blinding effect, the acupuncturist will also tap 2 guiding tubes at 2 sham points & immediately affix a pair of needles to the surface of the same points with adhesive tape, w
- Sham Acupuncture: Patients stratified based on cancer (breast cancer vs colorectal cancer). The patients will be randomly assigned to get sham acupuncture until the end of their chemo while following the same chemo dose reduction algorithm. No concomitant anti-neuropathy medication is allowed. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemo received in the past week. Record how much chemo received all together. Each week patient will have blood drawn (about 1 tsp) to check nerve growth factors levels.
  Sham Acupuncture using Park Sham placebo acupuncture device: Participants will get sham acupuncture until the end of chemo.
  Acupuncturist will insert Park Sham Devices, non-penetrating sham acupuncture device consisting of a retractable needle and an adhesive tube into the sham points, and then immediately apply 2 pieces of adhesive tape next to the needles. She will tap a mock plastic needle gui
- Total: Total of all reporting groups
Arm/Group | Standard Care | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 2 | 4 | 13 | 19
Age, Customized [Median (Full Range); unit: years] | 44 [42 to 45] | 50 [44 to 59] | 49 [33 to 65] | 49 [33 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 13 | 19
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Colorectal and Breast Cancer Patients in Each Arm Who Require Dose Reduction or Discontinuation Due to Chemotherapy-induced Peripheral Neuropathy.
Description: The main objective is to assess efficacy and safety of acupuncture using Seirin acupuncture needles in colorectal and breast cancer patients who developed chemotherapy-induced peripheral neuropathy while receiving adjuvant/neoadjuvant chemotherapy. Safety will be assessed by recording side effects from acupuncture treatment. Efficacy will be assessed by measuring the proportion of patients in each arm who are required to undergo dose reduction or discontinuation due to chemotherapy-induced peripheral neuropathy.
Time Frame: Week 12
Population: Zero participants analyzed due to early termination of study.
Groups:
- Acupuncture: Patients stratified based on cancer (breast cancer vs colorectal cancer). The patients will be randomly assigned to get acupuncture until the end of their chemo. Patient will complete a weekly questionnaire during the study to determine severity of nerve pain symptoms. Each week record the total amount of chemo received in the past week & all together. Each week patient will have blood drawn (about 1 tsp) to check nerve growth factors levels. All patients will follow the same chemo dose reduction algorithm. No concomitant anti-neuropathy medication allowed. In standard care arm, patients will not get additional therapy for CIPN. Acupuncture using Seirin® needles: Participants will get acupuncture weekly until the end of chemotherapy. Subjects will get acupuncture at documented acupoints. To improve blinding effect, acupuncturist will also tap 2 guiding tubes at 2 sham points & immediately affix a pair of needles to surface of the same points with adhesive tape, no needle insertion.
- Sham Acupuncture: Patients stratified based on cancer (breast vs colorectal). Patients to get sham acupuncture til the end of their chemo & following the same chemo dose reduction algorithm. No concomitant anti-neuropathy medication allowed. Pt complete a wkly questionnaire to determine severity of nerve pain symptoms. Each wk record the total amount of chemo in the past week & all together. Each wk patient have blood drawn (about 1 tsp) to check nerve growth factors levels. Sham Acupuncture using Park Sham placebo acupuncture device: Particip will get sham acupuncture til the end of chemo. Acupuncturist will insert Park Sham Devices, non-penetrating sham acupuncture device of a retractable needle & an adhesive tube into sham points &apply 2 pieces of adhesive tape next to needles; will tap a mock plastic needle guiding tube on surface of each of 8 true points in the arm & leg to produce some discernible sensation & then apply needle w/ piece of adhesive tape to dermal surface, w/out needle insertion.
Arm/Group | Standard Care | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Acupuncture: Patients stratified based on cancer (breast vs colorectal). Patients randomly assigned to get acupuncture until the end of their chemo. Patient will complete a weekly questionnaire to determine severity of nerve pain symptoms. Each week record the total amount of chemo received in the past week. Record how much chemotherapy received all together. Each week patient will have blood drawn (about 1 tsp) to check nerve growth factors levels. All patients will follow the same chemo dose reduction algorithm. No concomitant anti-neuropathy medication is allowed. In standard care arm, patients will not get additional therapy for CIPN.
  Acupuncture using Seirin® needles: Participants will receive acupuncture weekly until the end of chemotherapy.
  Subjects will get acupuncture at documented acupoints. To improve blinding effect, the acupuncturist will tap 2 guiding tubes at 2 sham points & affix a pair of needles to the surface of the same points with adhesive tape, without needle insertion.
- Sham Acupuncture: Patients stratified based on cancer (breast vs colorectal). The patients get sham acupuncture til the end of chemo with same chemo dose reduction algorithm. No concomitant anti-neuropathy medication is allowed. Patient complete a weekly questionnaire to determine severity of nerve pain symptoms. Weekly record total amount of chemo received in the past week & all together. Each week patient have blood drawn (about 1 tsp) to check nerve growth factors levels. Sham Acupuncture using Park Sham placebo acupuncture device: Particip will get sham acupuncture til the end of chemo. Acupuncturist will insert Park Sham Devices, non-penetrating sham acupuncture device consisting of a retractable needle & adhesive tube into the sham points, & then apply 2 pieces of adhesive tape next to needles. Will tap mock plastic needle guiding tube on the surface of each of 8 true points in arm & leg to produce sensation & apply a needle with piece of adhesive tape to dermal surface, no needle insertion.
Arm/Group | Standard Care | Acupuncture | Sham Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/13
Other Adverse Events (participants affected / at risk) | 0/2 | 3/4 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=2) | Acupuncture (N=4) | Sham Acupuncture (N=13)
rash, bruising & scabs (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) — rash on right arm near inner elbow, slight bruising on left top of foot below second toe, pin needle scabs, redness & bruising
swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) — swollen feet
visual impairment, numbness, trouble writing, loss of balance (General disorders) | 0 (0) | 1 (1) | 0 (0) — visual impairment, numbness, trouble writing, loss of balance

LIMITATIONS AND CAVEATS:
The PI left the institution before the end of the study; therefore the study was withdrawn in clinicaltrials.gov and IRB closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes